CLINICAL TRIAL: NCT02002962
Title: Radiofrequency Ablation Plus Botulinum Toxin Injection Versus Radiofrequency Ablation Only in Patients With Atrial Flutter to Prevent Post-procedural Atrial Fibrillation
Brief Title: Radiofrequency Ablation Plus Botulinum Toxin Injection Versus Radiofrequency Ablation Only in Patients With Atrial Flutter
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BT_AFL
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter | interventions — Radiofrequency Ablation; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA+BT injection (Active Comparator): Transseptal puncture is performed by used standard endovascular approach. Injection of the botulinum toxin is performed in main anatomical zones of ganglionated plexuses of left atrium using Myostar catheter (Biosense Webster).
  Interventions: Procedure: radiofrequency ablation; Drug: Botulinum Toxin Type A injection
- RFA (Active Comparator): Externally-irrigated tip (5-mm tip, Celsius Thermo-Cool, Biosense Webster, Diamond Bar, CA, USA). Temperature-controlled RF delivery was performed with a maximum power output of 50 W and temperature limit of 50 C. The catheter was irrigated using 0.9% saline infusion at a ﬂow rate of 20-40 mL/min during RF delivery and 2 mL/min between applications using a commercially available pump (Cool Flow, Biosense Webster).
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation
Drug: Botulinum Toxin Type A injection
  Arms: RFA+BT injection

SUMMARY:
The aim of this randomized study was to assess the effectiveness of endomyocardial botulinum toxin injection for preventing post-procedural atrial fibrillation in patients undergoing the radiofrequency ablation of atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECG documented paroxysmal or persistent AFL
* No prior documented history of AF
* Patient undergoing RFA of AFL.
* No indication (other than AFL) for continued anticoagulation with warfarin.
* No existing implantable cardiac device (pacemaker, defibrillator, cardiac resynchronization therapy device)

Exclusion Criteria:

* A history of atrial fibrillation
* Previous AF ablation procedure
* Congestive heart failure
* Left Ventricle ejection fraction less than 35%
* Unwillingness to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
number of paroxysms of atrial fibrillation | 1 year

SECONDARY OUTCOMES:
AF burden | 1 year
serious adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru